CLINICAL TRIAL: NCT04428762
Title: Glycemic Control and Quality of Life With i- Port Advance in Pediatric T1DM: Multi Center Crossover and Prospective Assessment
Brief Title: Glycemic Control and Quality of Life With i- Port Advance in Pediatric T1DM
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: we decided to change the protocol completely to an RCT.
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Collaborators: Sheba Medical Center (Other Government); Kaplan Medical Center (Other); Soroka University Medical Center (Other); Wolfson Medical Center (Other Government); Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 0100-18-ASF
Record Dates: First submitted 2019-07-03; First posted 2020-06-11 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-08

CONDITIONS: T1DM

STUDY DESIGN:
Intervention Model Description: This is a multi-center,2 parts study:
  the first part: randomized crossover study second part: prospective follow-up study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- I-Port use arm (Experimental)
  Interventions: Device: I-Port Advance use
- Regular injection arm (No Intervention)

INTERVENTIONS:
Device: I-Port Advance use — participants will apply I-port advance for 4 weeks and will inject all insulin through the port. follow up 3 months with/ without i-port.
  Arms: I-Port use arm

SUMMARY:
The incidence of T1DM in children, especially infants under 4 years of age, is increasing in the last decade. Not all patients are willing or able, from different reasons, to be treated with insulin pumps. This portion of patients' needs subcutaneous insulin injections, at lest 4 injections per day, sometimes up to 8 injections per day.

The recommended treatment is insulin injection before each carbohydrate content meal. Since each injection may lead to pain, many patients do not inject all recommended doses. The solution could be: eat with no bolus, or not to correct glucose level to retrain from pain sensation. I-Port use is able to address this issue by reducing the pain sensation accompanied with the injection. I-Port advance may give a technological solution to non-insulin pump T1DM pediatric patients.

There are no reports in the literature of the use of iport in children and youth. This information is essential since 95% of pediatric diabetes mellitus cases are insulin dependent and require multiple injections. Better balanced diabetes in childhood may prevent complications to long range and long-term diabetes therapy. Moreover, if discovered safe, the iport can be used also for other subcutaneously delivered medication in children, such as somtostatin analog, human growth hormone and clexane Study is designed as 2 parts. Initial part is a cross over design to compare between ipor use an injections regarding glucose in range, side effects and quality of life.

Second part is designed as prospective. To assess glycemic control with iport use or 3 months .

DETAILED DESCRIPTION:
study withdrawn Nor relevant

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with type 1 diabetes mellitus
2. Insulin injection ≥2 per day for at least a week.
3. Use of MDI insulin: Novorapid, Humalog or Apidra.
4. Ability and willingness to perform at least 3 daily self-measured plasma glucose profiles
5. Ability and willingness to adhere to the protocol. -

Exclusion Criteria:

1. Insulin pump use
2. Mix insulin use -

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
Life quality and satisfaction measures | 3 months from patient first enrollment
  Life quality measure before and after I-Port Advance use by questionnaire-delta of score
Adverse effect | 3 months from patient first enrollment
  Number of Adverse effect while using I-port-clinical

SECONDARY OUTCOMES:
Glycemic control evaluation | 3 months from patient first enrollment
  HbA1C% before and after 3 month use of I-port advance